CLINICAL TRIAL: NCT01638221
Title: Comparison of Patient Perceived Pain and Satisfaction Between Lightweight and Heavyweight Mesh for Laparoscopic Inguinal Hernia Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Adam Pentel, DO, general surgery resident, Ascension Health
Other Study IDs: ME10 0006
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- heavy weight mesh: Surgipro mesh is a heavier weighted mesh with less flexibility after surgery
- light weight mesh: UltraPro mesh is a lighter weighted mesh with theoretically less stiffness and more flexibility compared to heavier weighted meshes

SUMMARY:
This study will be comparing the patients overall satisfaction of two different meshes used in laparoscopic inguinal hernia repairs.

DETAILED DESCRIPTION:
This is a clinical trial comparing standard therapy in the use of either lightweight or heavy mesh for the repair of inguinal hernias. Both types of these meshes have been approved for surgical correction but subjective comparisons of patient overall satisfaction and perceived outcomes have not been measured. The investigators intend to measure certain subjective data in the form of a questionnaire will be issued to the patient preoperatively, one week, one month, six months, and one year after the surgery There is no recent literature comparing subjective data between two meshes called Ultra Pro and Surgi Pro. The biological effects of these meshes have identical properties as far as the healing process and inflammation as well as the low rate of infection. The main difference is the material that these meshes are composed of. The Ultra Pro is made of Prolene while the Surgi Pro is made of polypropylene.

The risks are not increased anymore than that for normal surgical complications. They each have the same post operative risks including bleeding, infection and pain, but the investigators are investigating a possible subjective difference between these two separate meshes that are currently used.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* unilateral side to be repaired
* no major abdominal surgery previously

Exclusion Criteria:

* under age 18
* bilateral repairs undertaken

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who are undergoing a unilateral repair of inguinal hernias laparoscopically
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
pain | 1 year
  Subjective pain scale rating post surgical

SECONDARY OUTCOMES:
return to activities of daily living | 1 year
  returning to their presurgical lifestyle

CONTACTS AND LOCATIONS:
Overall Officials: Adam P Pentel, DO, Principal Investigator — Ascension Health
Locations (1):
- GenesysRMC, Grand Blanc, Michigan, United States